CLINICAL TRIAL: NCT06494501
Title: The Prevent Coronary Artery Disease Trial
Acronym: PRECAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Valentin Fuster, Chairman Mount Sinai Fuster Heart Hospital, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-23-01528
Record Dates: First submitted 2024-06-23; First posted 2024-07-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inclisiran (Experimental): Participants in this arm will receive the study drug (inclisiran, for 5 years). Specific measures will be implemented to achieve the following goals: LDL-C <55 mg/dl; blood pressure <130/80 mmHg; and HbA1c <6.5%. Diet and lifestyle recommendations will be recommended to all patients as a first step. Follow-up will occur every 2 months until goals are achieved. If the goal is not achieved, the subsequent recommendation will be implemented. Pharmacologic treatment may be implemented as early as the first visit at the discretion of the physician.
  * Product Name: inclisiran
  * Active ingredient: inclisiran sodium
  * Dosage Form: Solution for Injection
  * Unit Dose Inclisiran sodium 300 mg/1.5 mL vial (equivalent to 284 mg inclisiran)
  * Route of Administration: SC use
  * Physical Description: Clear, colorless to pale yellow solution essentially free of particulates
  Interventions: Drug: Inclisiran
- Control Group (No Intervention): Participants in this group will receive guideline directed medical treatment, according to American Heart Association/American College of Cardiology guidelines. These recommendations will be provided to the primary care physicians to be followed, according to standards of care. Follow-up visits will occur every 6 months, although patients might be seen more often according to their provider´s criteria.

INTERVENTIONS:
Drug: Inclisiran — Subjects will be administered a single subcutaneous injection of 284 mg inclisiran for injection at predefined time points.
  Other Names: Leqvio
  Arms: Inclisiran

SUMMARY:
Despite increasing evidence that exposure to cardiovascular risk factors (CVRF) at an early age increases the prevalence of subclinical atherosclerosis and is associated with a greater risk of cardiovascular events later in life, there is a lack of randomized trial evidence to support primary prevention strategies in adults aged 30-50 years. The researchers have designed a randomized controlled trial to evaluate whether strict control of CVRF in young adults without known cardiovascular disease, will reduce the progression of total atherosclerosis burden, a surrogate endpoint for symptomatic cardiovascular disease, compared with usual care.

The researchers propose a randomized controlled trial enrolling 1,600 healthy young adults who meet the inclusion criteria and who do not meet any exclusion criteria. Eligible study participants will be randomized, in a 1:1 ratio, to either the intervention group (active treatment strategy) or to the control group (guideline-directed medical therapy). Randomization will be stratified by the presence or absence of atherosclerotic plaque in vascular ultrasound.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the most common cause of death in the world and contributes importantly to the majority of the world's deaths. Substantial data suggest that maintaining optimal population serum low density lipoprotein cholesterol (LDL-C), starting early in life, has the potential to lower the risk of incident ASCVD. However, this strategy of early initiation of LDL-C lowering therapies would represent a major paradigm shift from current guideline-based practice. Widespread acceptance and implementation of this approach in the medical community necessary to gain a population benefit will require a randomized clinical trial demonstrating benefit. Thus, the researchers will begin a trial, PRECAD, that evaluates LDL-C lowering in the early adult years through measurements of subclinical atherosclerosis.

The significance of subclinical atherosclerosis has been established in population-based studies. In a cohort of >4,000 subjects between 40-54 years, the Progression of Early Atherosclerosis (PESA) study showed that 63% of the asymptomatic participants presented subclinical atherosclerosis, and that it progresses with time. Subclinical atherosclerosis was associated with cardiovascular events along 10 years of follow-up in the CAFES-CAVE study. Similar findings were reported from the BioImage study in the HRP cohort have shown that presence of plaque, even in asymptomatic phases, improved risk reclassification and was independently associated with adverse cardiovascular events in long-term follow-up. Hence, demonstrating prevention of atherosclerosis progression is strongly suggestive of future clinical benefit.

LDL-C, even at levels currently considered normal, is independently associated with the presence and extent of early systemic atherosclerosis in the absence of major cardiovascular risk factors. These findings support more effective LDL-C lowering for primary prevention.

Research from multiple observational cohort studies has shown that risk of cardiovascular disease increases with increased exposure to elevated LDL-C, independent of other risk factors, in a concentration-dependent fashion. In the CARDIA study, which enrolled adults aged 18- 30 years with a median 16-year follow-up, incident cardiovascular disease risk increased as accumulation of exposure to LDL-C increased. Further, LDL-C level predicts progression of subclinical atherosclerosis measured by the PESA score, and subclinical atherosclerosis progression predicts CHD. For the composite event of all-cause death, nonfatal myocardial infarction, or nonfatal stroke, the updated event outcomes have the following distribution across PESA score categories: no disease (n=1,536), number of events = 10 (0.65%); focal (n=875), number of events = 8 (0.91%); intermediate (n=1,112), number of events = 13 (1.17%); generalized (n=547), number events = 13 (2.38%). These preliminary results, although unpublished, provide a rationale that higher PESA score portends a higher clinical event rate.

Under a different imaging score of atherosclerosis burden, a similar association between atherosclerosis burden and clinical event rate has also been observed in the preliminary (unpublished) data of the BioImage Study. The connection between the atherosclerosis burden and incident CHD offers a surrogate endpoint for CHD that will progress sooner, permitting a much shorter trial that will convincingly assess the primary prevention benefit of maintaining low LDL-C beginning early in adult life.

Strict diet and aggressive lifestyle changes are associated with LDL-C reduction, but adherence is generally poor. In the last year, the World Health Organization has included new strategies such as the polypill in its list of essential medicines, in response to the limitation that lack of adherence places on the management of patients, particularly in the setting of prevention.

Particularly difficult is to guarantee adherence in young populations due to the absence of risk awareness. Thus, new strategies should be implemented to guarantee adherence in these population subgroups. Inclisiran is a small interfering RNA administered twice-yearly (after the initial and 3-month doses) by a health care professional via subcutaneous injection that decreases production of proprotein convertase subtilisin-lexin type 9 (PCSK9) in the liver to low LDL-C levels. This treatment has been shown as a safe, effective, and well tolerated in a diverse population, and could represent a great opportunity to increase adherence in the setting of primary prevention.

A population requiring special attention are patients with familial hypercholesterolemia (FH). LDL-C is 2 times higher in patients with heterozygous FH, and 4-5 times higher in patients with homozygous familial hypercholesterolemia compared to the general population. Based on the high baseline LDL-C levels in FH patients, lowering of LDL-C may not be achieved with statins alone. Inclisiran has also been shown effective in adults with FH who are treated with maximally tolerated statin therapy with or without ezetimibe.

The hypothesis is that compared to usual care, maintaining LDL-C below 55 mg/dL, beginning in the early adult years (30-50 years), in addition to a strict control of other risk factors, will reduce progression of total atherosclerosis burden.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 30 to 50 years of age.
* No prior history of coronary artery disease, cerebrovascular disease or peripheral artery disease.
* Serum LDL-C > 1.8 mmol/l (70 mg/dl).
* Presence of subclinical atherosclerosis as assessed by 3DVUS or by the presence of coronary artery calcium (defined as coronary artery calcium score ≥25), independent of risk calculators; and/or high lifetime risk (≥30%) using the ASCVD calculator; and/or intermediate 10-year risk (≥7.5%) using the ASCVD calculator in the presence of 2 risk enhancers.

The presence of atherosclerotic plaque by 3DVUS will be defined according to the PESA study definitions14: plaque is defined as a focal protrusion into the arterial lumen of thickness >0.5 mm or >50% if the intima media thickness or intima media thickness >1.5 mm. CT scan for coronary artery calcium assessment will not be part of the protocol but will be used where available.

Risk enhancers are defined as15:

* Family history of premature atherosclerotic CVD
* Persistently elevated LDL-C ≥ 160 mg/dl
* Chronic kidney disease
* Metabolic syndrome
* Conditions specific to women (e.g. preeclampsia, premature menopause)
* Inflammatory diseases (especially rheumatoid arthritis, psoriasis, HIV)
* Ethnicity (e.g., South Asian ancestry)
* Persistently elevated triglycerides (≥175 mg/dl)
* Hs-CRP ≥2 mg/L
* Lp(a) levels >50 mg/dl
* apoB ≥130 mg/dl
* Ankle-brachial index <0.9

Exclusion Criteria:

Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the subject at significant risk (according to investigator's [or delegate] judgment) if he/she participates in the clinical study.

* An underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate) might interfere with interpretation of the clinical study results.
* Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least two methods of highly effective contraception (failure rate less than 1% per year) (e.g. combined oral contraceptives, barrier methods, approved contraceptive implant, long- term injectable contraception, or intrauterine device) for the entire duration of the study.
* Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 5 years.
* History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the three years prior to randomization
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in ALT, aspartate aminotransferase (AST), >3x the ULN, or total bilirubin >2x ULN at screening confirmed by a repeat abnormal measurement at least 1 week apart.
* Known contraindications to anti-lipid therapy
* Known history of alcohol and/or drug abuse within the last 5 years.
* Treatment with other investigational products or devices within 30 days or five half- lives of the screening visit, whichever is longer.
* Planned use of other investigational products or devices during the course of the study.
* Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:

  * Subjects who are unable to communicate or to cooperate with the investigator.
  * Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including subjects whose cooperation is doubtful due to drug abuse or alcohol dependency).
  * Unlikely to comply with the protocol requirements, instructions, and study- related restrictions (e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study).
  * Have any medical or surgical condition, which in the opinion of the investigator would put the subject at increased risk from participating in the study.
  * Persons directly involved in the conduct of the study.
* Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9.
* History of hypersensitivity to the study treatment or its excipients or to other siRNA drugs.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in atherosclerotic plaque burden from baseline | Baseline, 2.5 years and 5 years after randomization
  Change in atherosclerotic plaque burden at 2.5 years and the last year of follow up from baseline as measured by the 3D vascular ultrasound. Atherosclerotic plaque burden is amount of plaque in the arteries.

SECONDARY OUTCOMES:
Change in Number of participants with Cardiovascular Disease (CVD) | Baseline and 5 years after randomization
  Change in Number of participants with Cardiovascular Disease (CVD) at 5 years as compared to baseline. CVD includes myocardial infarction, stroke, revascularization), cardiovascular death and all cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Fuster Heart Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No